CLINICAL TRIAL: NCT05192629
Title: Prospective, Randomized, Double-blind, Double-dummy, Active-controlled, Phase 3 Clinical Trial Comparing the Safety and Efficacy of Intranasal Dexmedetomidine to Oral Midazolam as Premedication for Propofol Sedation in Pediatric Patients Undergoing Magnetic Resonance Imaging
Brief Title: Intranasal Dexmedetomidine Versus Oral Midazolam as Premedication for Propofol Sedation in Pediatric Patients Undergoing Magnetic Resonance Imaging
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, department of Anesthesiology, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUB-PED-MIDEX_MRI
Record Dates: First submitted 2021-12-28; First posted 2022-01-14 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: MRI; Pediatric Sedation; Midazolam; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be assessed in the preoperative anaesthesia consultation. If they meet the criteria for inclusion in our protocol, and have no exclusion criteria, the study will be explained to their parents (and to the child in simple language if they are old enough to understand). On the sedation day, randomisation is carried out by the clinical research unit of the H.U.D.E.R.F. The result of the randomisation is transmitted in opaque and sealed envelopes to the non-blinded members of the team who are responsible for preparing the premedications. Once prepared and anonymously labelled, the premedication is administered to the patient by the blinded nursing staff. The child is monitored for the next 30 minutes. Ten minutes before the examination, the child and his/her parents are taken to the induction room to meet the anesthesiologist who will take charge of the child.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Midazolam (Active Comparator): Administration of oral midazolam (0.25 mg/kg) as premedication before propofol-based sedation.
  The patient receives an oral premedication containing 0.125mL/kg of midazolam (which corresponds to a dosage of 0.25mg/kg of Ozalin® 2mg/ml, with a maximum of 20 mg). He/she also receives an intranasal spray containing matching placebo of dexmedetomidine (NaCl 0.9%). The volume administered corresponds to 0.02 mL/kg (which corresponds to a dosage of 2 mcg/kg of pure dexmedetomidine 100 mcg/mL in group D).
  Interventions: Drug: Midazolam
- Group Dexmedetomidine (Experimental): Administration of intranasal dexmedetomidine as premedication before propofol-based sedation.
  The patient receives an intranasal premedication containing 2 mcg/kg of dexmedetomidine. He/she also receives an oral solution containing matching placebo of midazolam (flavored-water prepared by the pharmacy). The volume administered corresponds to 0.125 mL/kg (which corresponds to a dosage of 0.25mg/kg of Ozalin® 2mg/mL, with a maximum of 20 mg or 10mL).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Premedication by intranasal dexmedetomidine
  Arms: Group Dexmedetomidine
Drug: Midazolam — Premedication by intranasal midazolam
  Arms: Group Midazolam

SUMMARY:
A magnetic resonance imaging (MRI) examination usually takes 30 to 45 minutes and requires the patient to remain perfectly still during the entire acquisition process to ensure quality. Children under 6 years of age are not very cooperative and sedation is required for this age group.

Currently, there are no specific recommendations for sedation for a paediatric MRI examination. In 2018, a retrospective study on the sedation protocol applied at Hôpital Universitaire des Enfants Reine Fabiola (H.U.D.E.R.F.) was conducted. In this protocol, premedication was done with oral midazolam and sedation with iterative boluses of propofol. This study concluded that the protocol in place was effective, but found that image acquisition during the procedure was interrupted in 25% of cases, largely due to involuntary movements of the child.

Preoperative stress can be emotionally traumatic for the child and may even extend beyond the perioperative period, hence the importance of premedication. For the most anxious children, non-pharmacological means of premedication are often not sufficient. Moreover, the literature shows that pharmacological premedication is useful in reducing parental separation anxiety and in facilitating induction of anaesthesia.

Midazolam is an effective premedication agent with some disadvantages (paradoxical reaction, low compliance of oral intake). Dexmedetomidine is a highly effective α-2 receptor agonist that can also be used as premedication according to the current literature. A report by the Pediatric Sedation Research Consortium (P.S.R.C.) shows that it has a safe profile and an incidence rate of serious adverse events of 0.36% in the paediatric population. Furthermore, administered intranasally, it is non-invasive, painless and has good bioavailability (over 80%).

The primary objective is to demonstrate the superiority of intranasal dexmedetomidine over oral midazolam as a premedication for bolus sedation of propofol in terms of the incidence of any event during the MRI procedure requiring temporary or permanent interruption of the examination.

The impact of dexmedetomidine on the amount of propofol administered and on the post-sedation period, the impact of external factors on the primary objective, the acceptance of intranasal premedication by the children and the quality of the MRI images will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, aged 6 months to 6 years,
* ASA score I to IV,
* Requiring standard magnetic resonance imaging due to clinical condition, regardless of underlying pathology,
* Sedation performed by an anesthesiologist,
* Written informed consent in accordance with the ICH-GCP and local legislation prior to trial entry.

Exclusion Criteria:

* Contraindications to MRI (cardiac pacemaker, neurostimulator, ferromagnetic implant),
* Sedation carried out by a non-anesthesiologist,
* Emergency MRI,
* Presence of head trauma,
* Presence of nasal congestion or upper respiratory tract infection on the day of sedation,
* Multiple procedures during the same sedation (operating room, evoked potentials, etc.),
* Children with pathologies requiring airway safety,
* Any known allergic or hypersensitivity reaction to dexmedetomidine,
* Any known allergic or hypersensitivity reaction to benzodiazepines,
* Concomitant use of negative chronotropes, as Digoxine,
* Patient known with chronic respiratory failure or myasthenia,
* Patient known with anatomical abnormality of the airway, lung disease or sleep apnea syndrome
* Patient with known cardiac rhythm abnormality or cardio-vascular disease,
* Patient with known hepatic disorder or chronic kidney disease,
* Patient with hypotension or bradycardia on the day of the examination,
* Patient with a BMI > 97th percentile (which corresponds to overweight, including obesity).

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of bradycardia | 6 hours
  Incidence of bradycardia (defined as a decrease of 2 standard deviations from normal for age, as described by the American Heart Association (AHA) in the Pediatric Advanced Life Support (PALS) manual, and which requires intervention by the anesthesiologist in charge of the patient to improve heart rate and cardiac output); expressed as percentage of patients
Hypotension | 6 hours
  Incidence of hypotension (defined as a systolic blood pressure below the 5th percentile for age, as described by the AHA in the PALS manual, and which requires intervention by the anesthesiologist in charge of the patient to improve blood pressure); expressed as percentage of patients
Desaturation | 6 hours
  Incidence of oxygen desaturation under 95% (defined as moderate if SpO2 is between 90 and 95%, severe if below 90%); expressed as percentage of patients
Movements | 6 hours
  Incidence of involuntary movements requiring intervention by the anesthesiologist in charge of the patient to deepen sedation; expressed as percentage of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote CJ, Wilson S; AMERICAN ACADEMY OF PEDIATRICS; AMERICAN ACADEMY OF PEDIATRIC DENTISTRY. Guidelines for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures: Update 2016. Pediatrics. 2016 Jul;138(1):e20161212. doi: 10.1542/peds.2016-1212. PMID 27354454
- [Background] Gutmann A, Pessenbacher K, Gschanes A, Eggenreich U, Wargenau M, Toller W. Propofol anesthesia in spontaneously breathing children undergoing magnetic resonance imaging: comparison of two propofol emulsions. Paediatr Anaesth. 2006 Mar;16(3):266-74. doi: 10.1111/j.1460-9592.2005.01777.x. PMID 16490090
- [Background] Jung SM. Drug selection for sedation and general anesthesia in children undergoing ambulatory magnetic resonance imaging. Yeungnam Univ J Med. 2020 Jul;37(3):159-168. doi: 10.12701/yujm.2020.00171. Epub 2020 Apr 17. PMID 32299181
- [Background] Yip P, Middleton P, Cyna AM, Carlyle AV. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006447. doi: 10.1002/14651858.CD006447.pub2. PMID 19588390
- [Background] Ghai B, Jain K, Saxena AK, Bhatia N, Sodhi KS. Comparison of oral midazolam with intranasal dexmedetomidine premedication for children undergoing CT imaging: a randomized, double-blind, and controlled study. Paediatr Anaesth. 2017 Jan;27(1):37-44. doi: 10.1111/pan.13010. Epub 2016 Oct 13. PMID 27734549
- [Background] Chorney JM, Kain ZN. Behavioral analysis of children's response to induction of anesthesia. Anesth Analg. 2009 Nov;109(5):1434-40. doi: 10.1213/ane.0b013e3181b412cf. Epub 2009 Aug 27. PMID 19713262
- [Background] Leroy PL, Costa LR, Emmanouil D, van Beukering A, Franck LS. Beyond the drugs: nonpharmacologic strategies to optimize procedural care in children. Curr Opin Anaesthesiol. 2016 Mar;29 Suppl 1:S1-13. doi: 10.1097/ACO.0000000000000312. PMID 26926330
- [Background] Sadeghi A, Khaleghnejad Tabari A, Mahdavi A, Salarian S, Razavi SS. Impact of parental presence during induction of anesthesia on anxiety level among pediatric patients and their parents: a randomized clinical trial. Neuropsychiatr Dis Treat. 2017 Feb 20;12:3237-3241. doi: 10.2147/NDT.S119208. eCollection 2017. PMID 28260897
- [Background] Wollin SR, Plummer JL, Owen H, Hawkins RM, Materazzo F. Predictors of preoperative anxiety in children. Anaesth Intensive Care. 2003 Feb;31(1):69-74. doi: 10.1177/0310057X0303100114. PMID 12635399
- [Background] Jun JH, Kim KN, Kim JY, Song SM. The effects of intranasal dexmedetomidine premedication in children: a systematic review and meta-analysis. Can J Anaesth. 2017 Sep;64(9):947-961. doi: 10.1007/s12630-017-0917-x. Epub 2017 Jun 21. PMID 28639236
- [Background] Sun Y, Lu Y, Huang Y, Jiang H. Is dexmedetomidine superior to midazolam as a premedication in children? A meta-analysis of randomized controlled trials. Paediatr Anaesth. 2014 Aug;24(8):863-74. doi: 10.1111/pan.12391. Epub 2014 Mar 26. PMID 24666837
- [Background] Talon MD, Woodson LC, Sherwood ER, Aarsland A, McRae L, Benham T. Intranasal dexmedetomidine premedication is comparable with midazolam in burn children undergoing reconstructive surgery. J Burn Care Res. 2009 Jul-Aug;30(4):599-605. doi: 10.1097/BCR.0b013e3181abff90. PMID 19506498
- [Background] Radhika KP, Sreejit MS, Ramadas KT. Efficacy of midazolam as oral premedication in children in comparison to triclofos sodium. Indian J Anaesth. 2016 Jun;60(6):415-9. doi: 10.4103/0019-5049.183389. PMID 27330204
- [Background] Mahmoud M, Barbi E, Mason KP. Dexmedetomidine: What's New for Pediatrics? A Narrative Review. J Clin Med. 2020 Aug 24;9(9):2724. doi: 10.3390/jcm9092724. PMID 32846947
- [Background] Petroz GC, Sikich N, James M, van Dyk H, Shafer SL, Schily M, Lerman J. A phase I, two-center study of the pharmacokinetics and pharmacodynamics of dexmedetomidine in children. Anesthesiology. 2006 Dec;105(6):1098-110. doi: 10.1097/00000542-200612000-00009. PMID 17122572
- [Background] Sriganesh K, Saini J, Theerth K, Venkataramaiah S. Airway Dimensions in Children with Neurological Disabilities During Dexmedetomidine and Propofol Sedation for Magnetic Resonance Imaging Study. Turk J Anaesthesiol Reanim. 2018 Jun;46(3):214-221. doi: 10.5152/TJAR.2017.48285. Epub 2017 Nov 27. PMID 30140518
- [Background] Berkenbosch JW. Options and Considerations for Procedural Sedation in Pediatric Imaging. Paediatr Drugs. 2015 Oct;17(5):385-99. doi: 10.1007/s40272-015-0140-6. PMID 26156106
- [Background] Anttila M, Penttila J, Helminen A, Vuorilehto L, Scheinin H. Bioavailability of dexmedetomidine after extravascular doses in healthy subjects. Br J Clin Pharmacol. 2003 Dec;56(6):691-3. doi: 10.1046/j.1365-2125.2003.01944.x. PMID 14616431
- [Background] Li BL, Zhang N, Huang JX, Qiu QQ, Tian H, Ni J, Song XR, Yuen VM, Irwin MG. A comparison of intranasal dexmedetomidine for sedation in children administered either by atomiser or by drops. Anaesthesia. 2016 May;71(5):522-8. doi: 10.1111/anae.13407. Epub 2016 Mar 3. PMID 26936022
- [Background] Mekitarian Filho E, Robinson F, de Carvalho WB, Gilio AE, Mason KP. Intranasal dexmedetomidine for sedation for pediatric computed tomography imaging. J Pediatr. 2015 May;166(5):1313-1315.e1. doi: 10.1016/j.jpeds.2015.01.036. Epub 2015 Mar 6. PMID 25748567
- [Background] van Hoorn CE, Flint RB, Skowno J, Davies P, Engelhardt T, Lalwani K, Olutoye O, Ista E, de Graaff JC. Off-label use of dexmedetomidine in paediatric anaesthesiology: an international survey of 791 (paediatric) anaesthesiologists. Eur J Clin Pharmacol. 2021 Apr;77(4):625-635. doi: 10.1007/s00228-020-03028-2. Epub 2020 Oct 29. PMID 33119787
- [Background] Kumar L, Kumar A, Panikkaveetil R, Vasu BK, Rajan S, Nair SG. Efficacy of intranasal dexmedetomidine versus oral midazolam for paediatric premedication. Indian J Anaesth. 2017 Feb;61(2):125-130. doi: 10.4103/0019-5049.199850. PMID 28250480
- [Background] Peng K, Wu SR, Ji FH, Li J. Premedication with dexmedetomidine in pediatric patients: a systematic review and meta-analysis. Clinics (Sao Paulo). 2014 Nov;69(11):777-86. doi: 10.6061/clinics/2014(11)12. PMID 25518037
- [Background] Kim HJ, Shin WJ, Park S, Ahn HS, Oh JH. The sedative effects of the intranasal administration of dexmedetomidine in children undergoing surgeries compared to other sedation methods: A systematic review and meta-analysis. J Clin Anesth. 2017 May;38:33-39. doi: 10.1016/j.jclinane.2017.01.014. Epub 2017 Jan 15. PMID 28372674
- [Background] Gupta A, Dalvi NP, Tendolkar BA. Comparison between intranasal dexmedetomidine and intranasal midazolam as premedication for brain magnetic resonance imaging in pediatric patients: A prospective randomized double blind trial. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):236-240. doi: 10.4103/joacp.JOACP_204_16. PMID 28781452
- [Background] Cho JE, Kim WO, Chang DJ, Choi EM, Oh SY, Kil HK. Titrated propofol induction vs. continuous infusion in children undergoing magnetic resonance imaging. Acta Anaesthesiol Scand. 2010 Apr;54(4):453-7. doi: 10.1111/j.1399-6576.2009.02169.x. Epub 2009 Nov 23. PMID 19930245
- [Background] Nagoshi M, Reddy S, Bell M, Cresencia A, Margolis R, Wetzel R, Ross P. Low-dose dexmedetomidine as an adjuvant to propofol infusion for children in MRI: A double-cohort study. Paediatr Anaesth. 2018 Jul;28(7):639-646. doi: 10.1111/pan.13400. Epub 2018 Jun 7. PMID 29882298
- [Background] Mason KP, Park RS, Sullivan CA, Lukovits K, Halpin EM, Imbrescia ST, Cavanaugh D, Prescilla R, Fox VL. The synergistic effect of dexmedetomidine on propofol for paediatric deep sedation: A randomised trial. Eur J Anaesthesiol. 2021 May 1;38(5):541-547. doi: 10.1097/EJA.0000000000001350. PMID 33009191
- [Background] Sulton C, McCracken C, Simon HK, Hebbar K, Reynolds J, Cravero J, Mallory M, Kamat P. Pediatric Procedural Sedation Using Dexmedetomidine: A Report From the Pediatric Sedation Research Consortium. Hosp Pediatr. 2016 Sep;6(9):536-44. doi: 10.1542/hpeds.2015-0280. Epub 2016 Aug 11. PMID 27516413
- [Background] Mason KP. Sedation trends in the 21st century: the transition to dexmedetomidine for radiological imaging studies. Paediatr Anaesth. 2010 Mar;20(3):265-72. doi: 10.1111/j.1460-9592.2009.03224.x. Epub 2009 Dec 10. PMID 20015137
- [Background] Rosen DA, Daume JT. Short duration large dose dexmedetomidine in a pediatric patient during procedural sedation. Anesth Analg. 2006 Jul;103(1):68-9, table of contents. doi: 10.1213/01.ane.0000216289.52261.5e. PMID 16790628
- [Background] Tu Y, Liang Y, Xiao Y, Lv J, Guan R, Xiao F, Xie Y, Xiao Q. Dexmedetomidine attenuates the neurotoxicity of propofol toward primary hippocampal neurons in vitro via Erk1/2/CREB/BDNF signaling pathways. Drug Des Devel Ther. 2019 Feb 19;13:695-706. doi: 10.2147/DDDT.S188436. eCollection 2019. PMID 30858699
- [Background] Bhatt M, Kennedy RM, Osmond MH, Krauss B, McAllister JD, Ansermino JM, Evered LM, Roback MG; Consensus Panel on Sedation Research of Pediatric Emergency Research Canada (PERC) and the Pediatric Emergency Care Applied Research Network (PECARN). Consensus-based recommendations for standardizing terminology and reporting adverse events for emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2009 Apr;53(4):426-435.e4. doi: 10.1016/j.annemergmed.2008.09.030. Epub 2008 Nov 20. PMID 19026467
- [Background] Malviya S, Voepel-Lewis T, Tait AR, Merkel S, Tremper K, Naughton N. Depth of sedation in children undergoing computed tomography: validity and reliability of the University of Michigan Sedation Scale (UMSS). Br J Anaesth. 2002 Feb;88(2):241-5. doi: 10.1093/bja/88.2.241. PMID 11878656
- [Derived] Wabelo ON, Schmartz D, Giancursio M, De Pooter F, Caruso G, Fils JF, Van der Linden P. Prospective, randomized, double-blind, double-dummy, active-controlled, phase 3 clinical trial comparing the safety and efficacy of intranasal dexmedetomidine to oral midazolam as premedication for propofol sedation in pediatric patients undergoing magnetic resonance imaging: the MIDEX MRI trial. Trials. 2023 Aug 11;24(1):518. doi: 10.1186/s13063-023-07529-0. PMID 37568242